CLINICAL TRIAL: NCT06318845
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Pharmacokinetic Drug-drug Interaction of DHP2302R1 and DHP2302R2 in Healthy Adult Volunteers
Brief Title: Phase 1 Study of DHP2302R1 and DHP2302R2 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daehwa Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2302CS-1
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence A (Experimental): DHP2302R1 75 mg once daily for 7 days, followed by 2 weeks of washout period; then DHP2302R2 50 mg once daily for 7 days, followed by 2 weeks of washout period; then DHP2302R1 75 mg+DHP2302R2 50 mg once daily for 7 days
  Interventions: Drug: DHP2302R1; Drug: DHP2302R2
- Seqeunce B (Experimental): DHP2302R1 75 mg once daily for 7 days, followed by 2 weeks of washout period; then DHP2302R1 75 mg+DHP2302R2 50 mg once daily for 7 days, followed by 2 weeks of washout period; then DHP2302R2 50 mg once daily for 7 days
  Interventions: Drug: DHP2302R1; Drug: DHP2302R2
- Sequence C (Experimental): DHP2302R2 50 mg once daily for 7 days, followed by 2 weeks of washout period; then DHP2302R1 75 mg+DHP2302R2 50 mg once daily for 7 days, followed by 2 weeks of washout period; then DHP2302R1 75 mg once daily for 7 days
  Interventions: Drug: DHP2302R1; Drug: DHP2302R2
- Sequence D (Experimental): DHP2302R2 50 mg once daily for 7 days, followed by 2 weeks of washout period; then DHP2302R1 75 mg once daily for 7 days, followed by 2 weeks of washout period; then DHP2302R1 75 mg+DHP2302R2 50 mg once daily for 7 days
  Interventions: Drug: DHP2302R1; Drug: DHP2302R2
- Seqeunce E (Experimental): DHP2302R1 75 mg+DHP2302R2 50 mg once daily for 7 days, followed by 2 weeks of washout period; then DHP2302R2 50 mg once daily for 7 days, followed by 2 weeks of washout period; then DHP2302R1 75 mg once daily for 7 days
  Interventions: Drug: DHP2302R1; Drug: DHP2302R2
- Seqeunce F (Experimental): DHP2302R1 75 mg+DHP2302R2 50 mg once daily for 7 days, followed by 2 weeks of washout period; then DHP2302R1 75 mg once daily for 7 days, followed by 2 weeks of washout period; then DHP2302R2 50 mg once daily for 7 days
  Interventions: Drug: DHP2302R1; Drug: DHP2302R2

INTERVENTIONS:
Drug: DHP2302R1 — 75 mg per dose, once daily
Drug: DHP2302R2 — 50 mg per dose, once daily

SUMMARY:
The purpose of this study is to investigate the safety and drug interaction of DHP2302R1 and DHP2302R2 when administered alone versus in combination in healthy South Korean adult participants.

DETAILED DESCRIPTION:
This is a phase 1 open-label, multiple doses, 6-sequence, 3-period, and crossover study to evaluate the safety and pharmacokinetic drug interaction following 7 days of DHP2302R1 75 mg and DHP2302R2 50 mg in healthy South Korean adult participants.

A total of 42 participants, 7 per 6 groups, will enroll in the study. The participants will take 7 days of DHP2302R1 75 mg, DHP2302R1 50 mg alone or in combination, and 2 weeks of washout period at each period.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult, age ≥ 19 years at the time of screening
2. Body weight ≥ 50.0 kg, with body mass index (BMI) ≥ 18.0 kg/m2 and ≤ 30.0 kg/m2 at the time of screening
3. A subject with no congenital, treatment-requiring chronic diseases, pathologic symptoms, or findings on internal medicine examination.
4. A subject determined to be suitable for the study as a result of clinical laboratory tests, vital signs, medical examination (physical examination), 12-lead electrocardiogram, and other tests set according to the characteristics of the investigational drug.
5. A subject voluntarily decided to participate and agreed in writing to comply with the subject compliance for the duration of the clinical trial.

Exclusion Criteria:

1. A subject with a current clinically significant liver, kidney, nervous, psychiatric, respiratory, endocrine, hematologic, tumor, genitourinary, cardiovascular, digestive, musculoskeletal, etc. diseases or history

   1. Kidney disorders
   2. Liver disorders
   3. Those with bleeding disorders (peptic ulcer, intracranial hemorrhage, hemophilia, digestive tract bleeding, urinary tract bleeding, hemorrhage, vitreous hemorrhage, etc.)
2. For women, pregnant women (Urine-HCG positive) or nursing mothers
3. A subject hypersensitivity or history of clinically significant hypersensitivity to clopidogrel, tegoprazan, or any component of the investigational drug, aspirin, or benzimidazole
4. A subject with a genetic condition such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption
5. A subject with a history of gastrointestinal disease (Crohn's disease, ulcers, acute or chronic pancreatitis, etc.) or gastrointestinal surgery (but not simple appendectomy or hernia surgery) that may affect the absorption of the investigational drug.
6. A subject with clinically significant findings on 12-lead electrocardiogram at screening, including the following findings

   1. QTc > 450 ms in men and QTc > 470 ms in women
   2. PR interval > 200 ms
   3. QRS duration > 120 ms
7. A subject with the following findings in clinical laboratory tests at the time of screening

   1. AST, ALT, ALP, γ-GT, and Bilirubin total > 2 times the upper limit of normal range in clinical laboratory tests for liver function evaluation
   2. Creatinine level in the blood exceeds the reference range or eGFR calculated by the CKD-EPI formula less than 60 mL/min/1.73 m2
   3. CPK > 2.5 times the upper limit of the normal range in clinical laboratory tests
8. A subject with a history of drug abuse or positive urine drug screen for drugs of abuse
9. A subject with systolic blood pressure ≥ 150 mm Hg or ≤ 90 mm Hg or diastolic blood pressure ≥ 100 mm Hg or ≤ 60 mm Hg and pulse ≤ 40 bpm or ≥ 100 bpm, which was measured in the sitting position after at least 3 minutes of rest, at the time of screening
10. A subject administered drugs that induce or inhibit drug-metabolizing enzymes, such as barbiturates, within 1 month before the first dose.
11. A subject with an unusual diet that may affect the absorption, distribution, metabolism, and excretion of the investigational drug or consume foods that may affect drug metabolism
12. A subject who received any specialty or herbal medications that may affect the properties of the investigational product, including cyclosporine, CYP2C19 inhibitors, atazanavir, nelfinavir, or rilpivirine-containing preparations within 2 weeks before the first dose, or any over-the-counter (OTC) or vitamin preparations within 10 days (however, if the medication does not affect the pharmacokinetic properties of the investigational product, the subject may participate in the study at the discretion of the investigator).
13. A subject who participated in and received treatment in another clinical trial within 6 months before the first dose (however, the termination criteria for participation in another clinical trial shall be the day following the last dose.)
14. A subject who donated whole blood within 2 months before the first dose, or component blood within 1 month, or received a blood transfusion within 1 month, or needed to must donate blood from written informed consent to the time of PSV.
15. A subject with consistent alcohol consumption (> 21 units/week, 1 unit=10 g=12.5 mL of pure alcohol) within 6 months before the first dose or unavailable to stop alcohol consumption from written informed consent to the time of PSV
16. A subject who smokes with an average daily cigarette consumption greater than 10 cigarettes within 3 months before the first dose and who is unable to quit smoking from 24 hours before the first dose at each time point until the time of the last blood draw.
17. A subject with consumption of or inability to abstain from grapefruit (grapefruit)-containing foods from 48 hours before the first dose until the time of PSV
18. A subject with consumption of or inability to abstain from caffeine-containing foods (coffee, green tea, black tea, carbonated beverages, coffee milk, tonic drinks, etc.
19. A subject who engaged in vigorous exercise that exceeds the level of their daily routine from 48 hours before the first dose to the time of PSV, or unavailable to abstain from vigorous exercise.
20. A subject or his/her spouse or partner who is planning to become pregnant from written informed consent until 2 weeks after the last dose of investigational product, or is not using a reliable method of contraception (e.g., contraceptive administration and implantation or intrauterine device, sterilization (vasectomy, tubal ligation, etc.), barrier method (combination of spermicide with condoms, contraceptive vaginal septum, vaginal sponge, or neck cap)).
21. A subject unsuitable for participation in the study by the investigator for any reason other than the above inclusion/exclusion criteria

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-05-07 (Actual)

PRIMARY OUTCOMES:
AUClast of DHP2302R1 and DHP2302R2 | At baseline (0 hours), administration day (Day 5 to Day 9) in each period
  Systemic exposure of DHP2302R1 and DHP2302R2
Cmax of DHP2302R1 and DHP2302R2 | At baseline (0 hours), administration day (Day 5 to Day 9) in each period
  Plasma concentrations of DHP2302R1 and DHP2302R2

SECONDARY OUTCOMES:
Tmax of DHP2302R1 and DHP2302R2 | At baseline (0 hours), administration day (Day 5 to Day 9) in each period
  Secondary pharmacokinetic parameters of DHP2302R1 and DHP2302R2
AUC0-48 of DHP2302R1 and DHP2302R2 | At baseline (0 hours), administration day (Day 5 to Day 9) in each period
  Secondary pharmacokinetic parameters of DHP2302R1 and DHP2302R2
AUCinf of DHP2302R1 and DHP2302R2 | At baseline (0 hours), administration day (Day 5 to Day 9) in each period
  Secondary pharmacokinetic parameters of DHP2302R1 and DHP2302R2
t1/2 of DHP2302R1 and DHP2302R2 | At baseline (0 hours), administration day (Day 5 to Day 9) in each period
  Secondary pharmacokinetic parameters of DHP2302R1 and DHP2302R2
CL/F of DHP2302R1 and DHP2302R2 | At baseline (0 hours), administration day (Day 5 to Day 9) in each period
  Secondary pharmacokinetic parameters of DHP2302R1 and DHP2302R2
Vz/F of DHP2302R1 and DHP2302R2 | At baseline (0 hours), administration day (Day 5 to Day 9) in each period
  Secondary pharmacokinetic parameters of DHP2302R1 and DHP2302R2

CONTACTS AND LOCATIONS:
Locations (1):
- H Plus Yangji Hospital, Seoul, Gwanak-gu, South Korea

IPD SHARING:
Plan to Share IPD: No